CLINICAL TRIAL: NCT02326389
Title: Exercise and Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Susan Mcgurk, Associate Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3636
Record Dates: First submitted 2014-12-18; First posted 2014-12-29 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Cognitive functioning
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Exercise; Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and Cognitive Remediation (Experimental): The exercise intervention is a 10-week program involving 40 minutes of aerobic exercise targeting 60-75% of maximum heart rate on 3 days each week, with an additional 5-minute stretching warm up and cool down. The experimental group will participate in the exercise intervention as well as cognitive remediation.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive Remediation
- Cognitive Remediation Only (Active Comparator): Participants will be engaged in 30 hours of computer-based cognitive exercises with a standardized, widely used software package (Cogpack, Version 7.0, Marker Software), shown to improve cognitive functioning in multiple studies. One-hour sessions will be conducted 3 times per week for 10 weeks.
  Interventions: Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention is a 10-week program involving 40 minutes of aerobic exercise targeting 60-75% of maximum heart rate on 3 days each week, with an additional 5-minute stretching warm up and cool down.
  Arms: Exercise and Cognitive Remediation
Behavioral: Cognitive Remediation — Participants will be engaged in 30 hours of computer-based cognitive exercises with a standardized, widely used software package (Cogpack, Version 7.0, Marker Software), shown to improve cognitive functioning in multiple studies. One-hour sessions will be conducted 3 times per week for 10 weeks.

SUMMARY:
The purpose of this study is to evaluate the potential benefits of combining cognitive remediation and exercise in improving cognitive functioning and response to psychiatric rehabilitation.

DETAILED DESCRIPTION:
Impaired cognitive functioning is a common feature of schizophrenia and other serious mental illnesses that is related to poorer psychosocial functioning and less benefit from psychiatric rehabilitation. Research shows that cognitive remediation for persons with serious mental illness improves cognitive functioning and response to psychiatric rehabilitation. There is also evidence that physical activity such as aerobic exercise confers a benefit to cognitive functioning in both clinical and general population samples. The cognitive benefit of exercise is hypothesized to be the result of enhanced brain-derived neurotrophic factor (BDNF; a protein that promotes plasticity, reduces degeneration, and stimulates nerve cell survival). However, the potential synergistic effects of cognitive remediation and exercise on cognitive functioning have not been investigated in persons with serious mental illness. This pilot randomized controlled trial will evaluate the impact of adding a peer run exercise program to a standardized cognitive remediation program on cognitive functioning in 30 people with schizophrenia, schizoaffective disorder or bipolar disorder. All study participants will receive a 10-week cognitive remediation program shown in previous research to improve cognitive functioning. One-half (N = 15) of the participants will also receive a peer-led exercise program designed to promote cardiovascular fitness. The primary research questions addressed are: 1) Does the addition of the exercise program to cognitive remediation lead to greater improvements in cognitive functioning than cognitive remediation alone?, and, 2) Are improvements in cognitive functioning mediated (explained) by exercise-induced increases in BDNF? The results of this pilot study will inform the design of a larger, more definitive trial to evaluate the potential benefits of combining cognitive remediation and exercise in improving cognitive functioning and response to psychiatric rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. a DSM-5 diagnosis of schizophrenia, schizoaffective disorder or bipolar disorder based on the Structured Diagnostic Interview for DSM-5;
2. no changes in prescribed psychotropic medication dosage or type for at least 1 month;
3. medical clearance from a physician to participate in the exercise program;
4. currently exhibiting a sedentary lifestyle, as defined by exercising less than 3 days/wk for at least 20 minutes each time;
5. no current active suicidal ideation; and 6) fluent in English.

Exclusion Criteria:

1. positive screen for a major neurocognitive disorder (as indicated by a score below 23 on the Folstein Mini Mental Exam or a positive score on the HELPS Brain Injury Screening using only cognitive items for "P" items);
2. DSM-5 diagnosis of substance use disorder other than nicotine or caffeine in the last 6 months, or bulimia within the last 6 months;
3. body mass index greater than 45; a BMI of 45 was selected as the upper limit in order to screen out individuals with Class III obesity who might be more prone to musculoskeletal injuries than individuals with a BMI at or less than 45; and
4. for women, currently pregnant, plans to be pregnant in the next year, or currently breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Change in Neurocognitive functioning | post- 10 week intervention and 2 weeks after end of intervention
  The neurocognitive outcome variables will be assessed at baseline, the week following the 10-week program, and 2 weeks later. Neurocognitive tests for primary outcome variables are from the MATRICS Neurocognition Committee for use with people with schizophrenia. These include tests of 1) attention and vigilance, 2) verbal working memory, 3) verbal learning, 4) visual learning, and 5) information processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Susan McGurk, PhD, Principal Investigator — Boston University; Michael Otto, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] McGurk SR, Otto MW, Fulford D, Cutler Z, Mulcahy LP, Talluri SS, Qiu WQ, Gan Q, Tran I, Turner L, DeTore NR, Zawacki SA, Khare C, Pillai A, Mueser KT. A randomized controlled trial of exercise on augmenting the effects of cognitive remediation in persons with severe mental illness. J Psychiatr Res. 2021 Jul;139:38-46. doi: 10.1016/j.jpsychires.2021.04.033. Epub 2021 May 13. PMID 34022474